CLINICAL TRIAL: NCT02461225
Title: A Double-blind, Placebo-controlled Randomized Evaluation of the Effect of the Erchonia® FX-635™ on Diabetic Peripheral Neuropathy Foot Pain Clinical Study Protocol
Brief Title: Study of Low Level Laser Therapy to Treat Diabetic Peripheral Neuropathy Foot Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC_DPN
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Erchonia® FX-635™ (Active Comparator): The Erchonia® FX-635™ is made up of 3 independent 17 milliWatts (mW), 635 nanometers (nm) red laser diodes mounted in scanner devices with flexible arms positioned equidistant from each other.
  Interventions: Device: Erchonia® FX-635™
- Placebo Laser (Placebo Comparator): The Placebo Laser has the same appearance as the Erchonia® FX-635™ but does not emit any therapeutic light.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia® FX-635™ — The Erchonia® FX-635™ is made up of 3 independent 17 mW, 635 nm red laser diodes that are applied for 15 minutes to each foot. The diodes are positioned around the foot such that each of the 3 laser lights is positioned between 3 and 4 inches away from, but directed toward: a) the top of the foot (dorsal aspect); b) the bottom of the foot (plantar aspect); and c) the posterior tibial nerve within the tarsal tunnel. The laser diodes laze each of these 3 areas for 15 minutes simultaneously. Each subject receives 12 total procedure administrations with the Erchonia® FX-635™ across the consecutive 6-week procedure administration phase, 2 procedure administrations per week, each procedure administration approximately evenly spaced.
  Arms: Erchonia® FX-635™
Device: Placebo Laser — The Placebo Laser has the same appearance as the Erchonia® FX-635™ but does not emit any therapeutic light. It is applied for 15 minutes to each foot. The diodes are positioned around the foot such that each of the 3 laser lights is positioned between 3 and 4 inches away from, but directed toward: a) the top of the foot (dorsal aspect); b) the bottom of the foot (plantar aspect); and c) the posterior tibial nerve within the tarsal tunnel. The laser diodes laze each of these 3 areas for 15 minutes simultaneously. Each subject receives 12 total procedure administrations with the Erchonia® FX-635™ across the consecutive 6-week procedure administration phase, 2 procedure administrations per week, each procedure administration approximately evenly spaced.
  Arms: Placebo Laser

SUMMARY:
The purpose of this study is to determine whether low level laser therapy is effective in the reduction of foot pain associated with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
It is the goal of the current double-blind, placebo-controlled study to evaluate the efficacy of the Erchonia FX-635 which emits (3) 635nm red diodes, for providing temporary reduction of foot pain associated with diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Existing clinical diagnosis of diabetes induced Peripheral Neuropathy documented by a suitably qualified and licensed medical professional
* Significant spontaneous foot pain that occurs approximately equally (comparably) bilaterally
* Significant spontaneous pain of 50 or greater on the 0-100 Visual Analog Scale (VAS) for the feet overall
* Foot pain is chronic, defined as having been ongoing for at least 3 months, bilaterally
* Stable anti-diabetic medication regimen for the prior 30 days or on no anti-diabetic medication regimen for the prior 30 days
* Willing and able to refrain from consuming any non-study over-the-counter and/or prescription medications or therapies for the relief of pain/inflammation throughout study participation
* Primary language is English.

Exclusion Criteria:

* No definitive clinical diagnosis of diabetes induced Peripheral Neuropathy or foot pain is undiagnosed, or diagnosed as being other than, or in addition to, diabetes induced Peripheral Neuropathy
* Foot pain is unilateral or notably different between the two feet
* Self-reported Degree of Pain rating on the Visual Analog Scale (VAS) pain scale is less than 50 for both feet overall
* Serious organ disease or other serious primary disease merger
* Diabetes ketosis, ketoacidosis or severe infection within the past 2 weeks
* Current, active chronic pain disease
* Cancer or treatment for cancer in the past 6 months
* Use of any analgesics, or an equivalent of over-the counter or prescription NSAIDs (nonsteroidal anti-inflammatory drugs) within 7 days prior to study initiation
* Use of any antidepressants within 30 days prior to study initiation
* Use of any of the following prescription medications within 30 days prior to study initiation: Neurontin; Lyrica; Tramadol; Opioid medicines such as Ultram and Ultracet
* Injections of local anesthetics such as lidocaine within the past 30 days
* Surgical intervention to treat diabetic peripheral neuropathy foot pain, including implantation of a pain relief device
* Active infection, wound or other external trauma to the treatment areas
* Medical, physical, or other contraindications for, or sensitivity to, light therapy
* Pregnant, breast feeding, or planning pregnancy prior to the end of study participation
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years
* Developmental disability or cognitive impairment that in the opinion of the investigator would preclude adequate comprehension of the consent form and/or ability to record study measurements
* Involvement in litigation/receiving disability benefits related to the parameters of the study
* Participation in other research in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Zang, DPN, Principal Investigator
Locations (2):
- Arizona Institute of Footcare Physicians, Mesa, Arizona, United States
- Midleton Foot Clinic, Midleton, Co. Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia® FX-635™ | Placebo Laser
Started | 19 | 11
Completed | 19 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erchonia® FX-635™ | Placebo Laser | Total
Number analyzed (Participants) | 19 | 11 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.83 (13.19) | 53.45 (11.26) | 51.24 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 13 | 7 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Ireland | 19 | 11 | 30
Visual Analog Scale Pain Rating [Mean (Standard Deviation); unit: units on a scale] — The Visual Analog Scale assesses the level or degree of pain, from 0 to 100. It is a horizontal line labeled on the left '0: no pain at all' and on the right by the label '100: worst pain imaginable'. The subject marks a location on the 0-100 line that appears to represent any level of pain he or she is experiencing at that time. This marking is measured with a 0 to 100 mm ruler and the number recorded. A lower Visual Analog Scale pain score from baseline to study endpoint represents a better outcome, whereas a higher score from baseline to study endpoint represents a worse outcome.
  units on a scale | 68.89 (12.49) | 65.91 (10.69) | 67.88 (11.99)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 30% or Greater Change in Pain Rating on the Visual Analog Scale (VAS)
Description: The Visual Analog Scale (VAS) from baseline to endpoint (6 weeks) measurement is calculated for each subject. Individual subject success is defined as a 30% or greater change in VAS pain scores across the evaluation period. A negative (-) percent change indicates a decrease in pain level and is positive for individual subject success. A lower Visual Analog Scale pain score from baseline to study endpoint represents a better outcome, whereas a higher score from baseline to study endpoint represents a worse outcome.
  For the primary study outcome, the overall study success is defined as a 35% or greater difference between the proportion (number) of individual successes in each treatment group.
Time Frame: Baseline and 6 weeks
Measure: Number; unit: participants
Arm/Group | Erchonia® FX-635™ | Placebo Laser
Number analyzed (Participants) | 19 | 11
participants | 18 | 4
Statistical Analysis 1: Comparison: Erchonia® FX-635™ vs Placebo Laser; Test type: Superiority; p < .0005, Fisher Exact

2. Secondary Outcome: Change in Pain Rating on the Visual Analog Scale (VAS)
Description: The Visual Analog Scale (VAS) assesses level or degree of pain. It is a horizontal line anchored on the left by the label '0: no pain at all' and on the right by the label '100: worst pain imaginable'. The subject marks a location on the 0-100 line that appears to represent any level of pain he or she is experiencing at that time. This marking is measured with a 0 to 100 mm ruler and the number recorded. A lower Visual Analog Scale pain score from baseline to study endpoint represents a better outcome, whereas a higher score from baseline to study endpoint represents a worse outcome.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erchonia® FX-635™ | Placebo Laser
Number analyzed (Participants) | 19 | 11
score on a scale | -60.97 (23.28) | -9.09 (34.06)
Statistical Analysis 1: Comparison: Erchonia® FX-635™ vs Placebo Laser; Test type: Superiority; p < 0.0001, ANOVA

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Erchonia® FX-635™ | Placebo Laser
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/11
Other Adverse Events (participants affected / at risk) | 0/19 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-01-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT02461225/Prot_SAP_ICF_001.pdf